CLINICAL TRIAL: NCT02603809
Title: A Multi-center, Double-blind, Double-dummy, Randomized, Placebo- and Active-reference, Parallel Group, Phase 2, Dose-finding Study With ACT-132577 in Subjects With Essential Hypertension (Grade 1 and 2).
Brief Title: Dose-finding Study With ACT-132577 (Aprocitentan) in Participants With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-080A201
Record Dates: First submitted 2015-11-09; First posted 2015-11-13 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — aprocitentan; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): After a 4 to 6-week single-blind placebo run-in period, participants will be randomized to received placebo orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
  Interventions: Drug: Placebo
- Aprocitentan 5 mg (Experimental): After a 4 to 6-week single-blind placebo run-in period, participants will be randomized to received aprocitentan orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
  Interventions: Drug: Aprocitentan 5 mg
- Aprocitentan 10 mg (Experimental): After a 4 to 6-week single-blind placebo run-in period, participants will be randomized to received aprocitentan 10 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
  Interventions: Drug: Aprocitentan 10 mg
- Aprocitentan 25 mg (Experimental): After a 4 to 6-week single-blind placebo run-in period, participants will be randomized to received aprocitentan 25 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
  Interventions: Drug: Aprocitentan 25 mg
- Aprocitentan 50 mg (Experimental): After a 4 to 6-week single-blind placebo run-in period, participants will be randomized to received aprocitentan 50 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
  Interventions: Drug: Aprocitentan 50 mg
- Lisinopril 20 mg (Active Comparator): After a 4 to 6-week single-blind placebo run-in period, participants will be randomized to received lisinopril 20 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
  Interventions: Drug: Lisinopril 20 mg

INTERVENTIONS:
Drug: Aprocitentan 5 mg — One capsule of 5 mg aprocitentan, orally, once daily in the morning for 8 weeks, along with placebo capsule matching lisinopril.
  Other Names: ACT-132577
  Arms: Aprocitentan 5 mg
Drug: Aprocitentan 10 mg — Two capsules of 5 mg aprocitentan, orally, once daily in the morning for 8 weeks.
  Other Names: ACT-132577
  Arms: Aprocitentan 10 mg
Drug: Aprocitentan 25 mg — One capsule of 25 mg aprocitentan, orally, once daily in the morning for 8 weeks, along with placebo capsule matching lisinopril.
  Other Names: ACT-132577
  Arms: Aprocitentan 25 mg
Drug: Aprocitentan 50 mg — One capsule of 50 mg aprocitentan, orally, once daily in the morning for 8 weeks, along with placebo capsule matching lisinopril.
  Other Names: ACT-132577
  Arms: Aprocitentan 50 mg
Drug: Lisinopril 20 mg — One capsule of 20 mg lisinopril, orally, once daily in the morning for 8 weeks, along with placebo capsule matching aprocitentan
  Arms: Lisinopril 20 mg
Drug: Placebo — One capsule each of placebo matching aprocitentan and placebo matching lisinopril orally, once daily in the morning for 8 weeks.
  Arms: Placebo

SUMMARY:
The main objective will be to evaluate the dose-response of ACT-132577 (aprocitentan) on diastolic blood pressure (DBP) in participants with grade 1 or 2 essential hypertension.

Secondary objectives will be to evaluate the dose-response of ACT-132577 on: systolic blood pressure (SBP); control and response rate of blood pressure; 24-hour ambulatory blood pressure monitoring (ABPM) and to evaluate the safety and tolerability of a once daily oral regimen of 4 doses of ACT-132577.

DETAILED DESCRIPTION:
Participation in the study is planned to last up to 18 weeks. A single-blind placebo run-in period of 4 to 6 weeks after which participants will be randomized into a double-blind treatment period of 8 weeks and a washout and follow-up period ending with an end-of-study visit approximately 12 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* No contra-indication to stop (according to label) anti-hypertensive treatment(s) at screening
* Mild-to-moderate essential hypertension with or without ongoing anti-hypertensive treatment(s):

  -- Mean (of 5 measurements) sitting diastolic blood pressure (SiDBP) ≥ 90 to < 110 mmHg measured by office blood pressure measurements (OBPM).
* Women of childbearing potential must have a negative pregnancy test and use of reliable methods of contraception

Exclusion Criteria:

* Severe hypertension (grade 3): mean sitting systolic/diastolic BP (SiSBP/SiDBP; measured by OBPM) ≥ 180/110 mmHg, respectively.
* Secondary hypertension
* Known hypertensive retinopathy greater than Keith-Wagener Grade 2
* Myocardial infarction, percutaneous transluminal coronary angioplasty, or coronary artery bypass graft within 12 months prior to randomization
* Unstable angina within 6 months prior to randomization
* Heart failure New York Heart Association class III and IV
* Valvular defects (such as severe aortic or mitral valve disease) and/or hemodynamically relevant rhythm disturbances
* Clinical evidence of cerebrovascular insufficiency or a cerebrovascular accident within 6 months prior to randomization.
* Subjects working night shifts
* Body mass index < 20 kg/m2 or > 40 kg/m2
* Treatment with any medication which may affect BP (e.g., treatment of psychiatric diseases, ophthalmic preparations)
* Treatment with strong cytochrome P450 3A4 (CYP3A4) isoenzyme inhibitors or inducers
* Treatment with guanethidine and/or mineralocorticoid receptor antagonists within 1 month prior to Screening (Visit 1)
* Treatment with another investigational treatment within 1 month prior to Screening (Visit 1)
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1659 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ClinicalTrials, Study Director — Idorsia Pharmaceuticals
Locations (89):
- United States (73):
  - Appalachian Cardiovascular Associates, Fort Payne, Alabama
  - Radiant Research Inc, Chandler, Arizona
  - Warner Family Practice / Radiant Research Inc, Chandler, Arizona
  - Phoenix Medical Research Institute LLC, Peoria, Arizona
  - Advanced Arizona Clinical Research, Tucson, Arizona
  - Noble Clinical Research LLC, Tucson, Arizona
  - Desert Sun Clinical Research LLc, Tucson, Arizona
  - Advanced Research Center Inc, Anaheim, California
  - Med Center, Carmichael, California
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Clinical Trials Research, Lincoln, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Entertainment Medical Group Inc, Los Angeles, California
  - Artemis institute for Clinical Research, San Diego, California
  - Memorial Research Medical Clinic / Orange County Research Center, Tustin, California
  - Empire Clinical Research, Upland, California
  - Clinical Research Consulting LLC, Milford, Connecticut
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Alfieri Cardiology, Wilmington, Delaware
  - ACRC - Cardiology, Atlantis, Florida
  - Innovative Research of West Florida INC, Clearwater, Florida
  - Avail Clinical Research LLC, DeLand, Florida
  - Alan Graff, MD, PA, Fort Lauderdale, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Canvas Clinical Research, LLC, Lake Worth, Florida
  - LCC Medical Research Institute, Miami, Florida
  - Allied Biomedical Research Institute, INC, Miami, Florida
  - Southeast Regional Research Group, Savannah, Georgia
  - Community Clin Res CTR, Anderson, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Heartland Research Associated LLC, Newton, Kansas
  - Heartland Research Associates LLC, Wichita, Kansas
  - Avant Research Associates, LLC, Crowley, Louisiana
  - Best Clinical Trials LLC, New Orleans, Louisiana
  - New Orleans Center for Clinical Research - Nola, New Orleans, Louisiana
  - Clinsite LLC, Ann Arbor, Michigan
  - Primecare Research Associates, LLC, Florissant, Missouri
  - Clinical Research Advantage, Inc. / Diagnostic Center Of Medicine - Durango, Las Vegas, Nevada
  - Premier Research, Trenton, New Jersey
  - Rochester Clinical Research Inc., Rochester, New York
  - Metrolina Internal Medicine/Internal Medicine Research, Charlotte, North Carolina
  - Pharmquest LLC, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Sterling Research Group Ltd., Cincinnati, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Aventiv Research Inc., Dublin, Ohio
  - Oklahoma City Clinic - Edmond / Radiant Research Inc, Edmond, Oklahoma
  - Clinical Research Advantage, Inc. / Oklahoma City Clinic - Midwest City, Midwest City, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Detweiler Family Medicine and Associates PC, Lansdale, Pennsylvania
  - Suburban Research Center, Media, Pennsylvania
  - Degarmo Institute of Medical Research, Greer, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - Tekton Research Inc, Austin, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Trinity Hypertension & Metabolic Research Institute, Carrollton, Texas
  - Family Medicine Associates of Texas - ACRC Trials, Carrollton, Texas
  - Coastal Bend Clinical Research, Corpus Christi, Texas
  - TR - Global Medical Research, DeSoto, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - Avant Research Associates LLC, Port Arthur, Texas
  - Texas Diabetes & Endocrinology, Round Rock, Texas
  - Radiant Research Inc, San Antonio, Texas
  - Bandera Family Health Care, San Antonio, Texas
  - Wasatch Clinical Research LLC, Salt Lake City, Utah
  - Health Research of Hampton Roads, Newport News, Virginia
  - National Clinical Research Inc, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (7):
  - Manna Research - Vancouver, Vancouver, British Columbia
  - Canadian Phase Onwards Inc, Toronto, Ontario
  - Manna Research - Toronto, Toronto, Ontario
  - Manna Research - Levis, Lévis, Quebec
  - Diex Recherche Montreal Inc, Montreal, Quebec
  - Manna Research - Pointe Claire, Pointe-Claire, Quebec
  - Diex Reserach Sherbrooke Inc, Sherbrooke, Quebec
- Israel (7):
  - Cardiology Department Barzilai, Ashkelon
  - Soroka University Hospital - Hypertension Unit, Beersheba
  - The Hyper Unit, Edith Wolfson Medical Center, Holon
  - Hypertension Treatment Center, Internal Dep, Hadassah, Jerusalem
  - Hypertension And Nephrology Department, Meir Medical Center, Kefar Sava
  - Clinical Research Unit Kaplan Medical Center, Rehovot
  - Internal Med Department A, Ziv Medical Center, Safed
- Puerto Rico (2):
  - Advanced Medical Concepts, PSC, Cidra
  - Research & Cardiovascular Corp., Ponce

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verweij P, Danaietash P, Flamion B, Menard J, Bellet M. Randomized Dose-Response Study of the New Dual Endothelin Receptor Antagonist Aprocitentan in Hypertension. Hypertension. 2020 Apr;75(4):956-965. doi: 10.1161/HYPERTENSIONAHA.119.14504. Epub 2020 Feb 17. PMID 32063059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 99 sites in 3 countries. Of the 1659 participants that signed the informed consent 996 entered the run-in period (i.e. 663 participants were screening failures: 651 failed to meet the eligibility criteria to enter the run-in period, 6 withdrew and 6 did not enter the run-in period for other reasons).
Pre-assignment Details: Of the 996 participants enrolled into the run-in period, a total 992 participants received at least one dose of the single-blind placebo. Of these 992 participants 502 were considered run-in failures (390 failing to meet randomization criteria, 57 withdrew consent and 55 left for other reasons) and 490 participants were randomized into the study.
Groups:
- Placebo: After a 4 to 6-week single-blind placebo run-in period, participants received placebo orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Aprocitentan 5 mg: After a 4 to 6-week single-blind placebo run-in period, participants received 5 mg aprocitentan orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Aprocitentan 10 mg: After a 4 to 6-week single-blind placebo run-in period, participants received aprocitentan 10 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Aprocitentan 25 mg: After a 4 to 6-week single-blind placebo run-in period, participants received aprocitentan 25 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Aprocitentan 50 mg: After a 4 to 6-week single-blind placebo run-in period, participants received aprocitentan 50 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Lisinopril 20 mg: After a 4 to 6-week single-blind placebo run-in period, participants received lisinopril 20 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
Period: Overall Study
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
Started | 82 | 82 | 82 | 82 | 81 | 81
Per-protocol Set | 67 | 68 | 71 | 67 | 68 | 69
Modified Per-Protocol Set | 66 (One participant had out of analysis window blood pressure measurements.) | 68 | 71 | 67 | 68 | 69
Completed Study (Participants that completed the 30-day follow-up telephone call / visit (i.e., End-of-Study).) | 75 | 79 | 79 | 76 | 78 | 75
Completed (Participants that completed the 8-week treatment period.) | 70 | 74 | 75 | 70 | 70 | 71
Not Completed | 12 | 8 | 7 | 12 | 11 | 10
Not completed — Withdrawal by Subject | 4 | 1 | 2 | 3 | 3 | 4
Not completed — Lost to Follow-up | 2 | 3 | 1 | 4 | 2 | 2
Not completed — Pre-specified discontinuation criteria | 3 | 3 | 2 | 2 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Adverse Event | 3 | 0 | 2 | 2 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (N=490), i.e. all participants randomized.
Groups:
- Placebo: Participants randomized to placebo treatment for 8 weeks.
- Aprocitentan 5 mg: Participants randomized to 5 mg aprocitentan treatment for 8 weeks.
- Aprocitentan 10 mg: Participants randomized to 10 mg aprocitentan treatment for 8 weeks.
- Aprocitentan 25 mg: Participants randomized to 25 mg aprocitentan treatment for 8 weeks.
- Aprocitentan 50 mg: Participants randomized to 50 mg aprocitentan treatment for 8 weeks.
- Lisinopril 20 mg: Participants randomized to 20 mg lisinopril treatment for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg | Total
Number analyzed (Participants) | 82 | 82 | 82 | 82 | 81 | 81 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Per Protocol Set (PPS, N=410) 8 weeks in the double-blind period, and no major protocol deviation.
  In the placebo group, one participant had out of analysis window blood pressure measurement. This participant was part of the PPS but not part of the modified Per Protocol Set (N=409).
  years
    Full Analysis Set | 53.5 (9.1) | 54.1 (8.5) | 55.3 (9.8) | 55.1 (10.0) | 54.2 (9.3) | 56.0 (9.0) | 54.7 (9.3)
    Per Protocol Set: number analyzed (Participants) | 67 | 68 | 71 | 67 | 68 | 69 | 410
    Per Protocol Set | 53.9 (9.1) | 55.0 (8.5) | 55.8 (9.5) | 55.7 (9.8) | 54.0 (9.4) | 56.1 (9.4) | 55.1 (9.3)
    modified Per Protocol Set: number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69 | 409
    modified Per Protocol Set | 54.0 (9.1) | 55.0 (8.5) | 55.8 (9.5) | 55.7 (9.8) | 54.0 (9.4) | 56.1 (9.4) | 55.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Per Protocol Set (PPS, N=410) 8 weeks in the double-blind period, and no major protocol deviation.
  In the placebo group, one participant had out of analysis window blood pressure measurement. This participant was part of the PPS but not part of the modified Per Protocol Set (N=409).
  Participants
    Full Analysis Set: Female | 27 | 34 | 31 | 37 | 28 | 36 | 193
    Full Analysis Set: Male | 55 | 48 | 51 | 45 | 53 | 45 | 297
    Per Protocol Set: number analyzed (Participants) | 67 | 68 | 71 | 67 | 68 | 69 | 410
    Per Protocol Set: Female | 22 | 27 | 26 | 30 | 24 | 31 | 160
    Per Protocol Set: Male | 45 | 41 | 45 | 37 | 44 | 38 | 250
    modified Per Protocol Set: number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69 | 409
    modified Per Protocol Set: Female | 22 | 27 | 26 | 30 | 24 | 31 | 160
    modified Per Protocol Set: Male | 44 | 41 | 45 | 37 | 44 | 38 | 249
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per Protocol Set (PPS, N=410) 8 weeks in the double-blind period, and no major protocol deviation.
  Participants
    Full Analysis Set: Hispanic or Latino | 23 | 26 | 31 | 27 | 28 | 26 | 161
    Full Analysis Set: Not Hispanic or Latino | 59 | 56 | 51 | 55 | 53 | 55 | 329
    Full Analysis Set: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Per Protocol Set: number analyzed (Participants) | 67 | 68 | 71 | 67 | 68 | 69 | 410
    Per Protocol Set: Hispanic or Latino | 19 | 22 | 28 | 24 | 25 | 23 | 141
    Per Protocol Set: Not Hispanic or Latino | 48 | 46 | 43 | 43 | 43 | 46 | 269
    Per Protocol Set: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per Protocol Set (PPS, N=410) 8 weeks in the double-blind period, and no major protocol deviation.
  Participants
    Full Analysis Set: American Indian or Alaska Native | 1 | 0 | 2 | 1 | 0 | 0 | 4
    Full Analysis Set: Asian | 2 | 0 | 1 | 0 | 0 | 2 | 5
    Full Analysis Set: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Full Analysis Set: Black or African American | 31 | 28 | 26 | 35 | 26 | 32 | 178
    Full Analysis Set: White | 48 | 54 | 53 | 46 | 55 | 46 | 302
    Full Analysis Set: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Full Analysis Set: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Per Protocol Set: number analyzed (Participants) | 67 | 68 | 71 | 67 | 68 | 69 | 410
    Per Protocol Set: American Indian or Alaska Native | 0 | 0 | 2 | 1 | 0 | 0 | 3
    Per Protocol Set: Asian | 1 | 0 | 1 | 0 | 0 | 1 | 3
    Per Protocol Set: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Per Protocol Set: Black or African American | 26 | 22 | 19 | 26 | 21 | 26 | 140
    Per Protocol Set: White | 40 | 46 | 49 | 40 | 47 | 41 | 263
    Per Protocol Set: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Per Protocol Set: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 1 | 6 | 4 | 2 | 5 | 21
  United States | 75 | 75 | 74 | 73 | 75 | 71 | 443
  Israel | 4 | 6 | 2 | 5 | 4 | 5 | 26
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Per Protocol Set (PPS, N=410) 8 weeks in the double-blind period, and no major protocol deviation.
  In the placebo group, one participant had out of analysis window blood pressure measurement. This participant was part of the PPS but not part of the modified Per Protocol Set (N=409).
  kilograms
    Full Analysis Set | 92.0 (18.9) | 88.6 (16.9) | 90.1 (18.3) | 91.1 (16.9) | 87.6 (15.8) | 87.0 (17.2) | 89.4 (17.37)
    Per Protocol Set: number analyzed (Participants) | 67 | 68 | 71 | 67 | 68 | 69 | 410
    Per Protocol Set | 91.0 (19.2) | 88.3 (17.6) | 89.3 (19.0) | 91.7 (18.1) | 87.1 (15.8) | 86.5 (16.0) | 89.0 (17.7)
    modified Per Protocol Set: number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69 | 409
    modified Per Protocol Set | 90.6 (19.0) | 88.3 (17.6) | 89.3 (19.0) | 91.7 (18.1) | 87.1 (15.8) | 86.5 (16.0) | 89.0 (17.7)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] — Population: Per Protocol Set (PPS, N=410) 8 weeks in the double-blind period, and no major protocol deviation.
  In the placebo group, one participant had out of analysis window blood pressure measurement. This participant was part of the PPS but not part of the modified Per Protocol Set (N=409).
  kilograms per square meter
    Full Analysis Set | 30.6 (5.07) | 30.1 (4.56) | 30.8 (4.52) | 31.0 (4.16) | 30.2 (4.55) | 30.4 (4.59) | 30.5 (4.57)
    Per Protocol Set: number analyzed (Participants) | 67 | 68 | 71 | 67 | 68 | 69 | 410
    Per Protocol Set | 30.1 (5.1) | 29.8 (4.5) | 30.4 (4.6) | 31.0 (4.3) | 30.3 (4.7) | 30.4 (4.6) | 30.3 (4.6)
    modified Per Protocol Set: number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69 | 409
    modified Per Protocol Set | 30.1 (5.1) | 29.8 (4.5) | 30.4 (4.6) | 31.0 (4.3) | 30.3 (4.7) | 30.4 (4.6) | 30.3 (4.6)
Duration of essential hypertension at screening [Mean (Standard Deviation); unit: years] — Population: Per Protocol Set (PPS, N=410) 8 weeks in the double-blind period, and no major protocol deviation.
  years
    Full Analysis Set | 9.13 (8.72) | 8.12 (8.25) | 10.48 (10.18) | 9.56 (8.97) | 10.60 (9.95) | 11.79 (10.47) | 9.94 (9.48)
    Per Protocol Set: number analyzed (Participants) | 67 | 68 | 71 | 67 | 68 | 69 | 410
    Per Protocol Set | 9.24 (8.93) | 8.38 (8.62) | 10.6 (10.51) | 9.19 (8.61) | 10.35 (10.07) | 12.53 (10.88) | 10.06 (9.7)
Antihypertensive treatment at screening [Number; unit: participants] — Population: Per Protocol Set (PPS, N=410) 8 weeks in the double-blind period, and no major protocol deviation.
  In the placebo group, one participant had out of analysis window blood pressure measurement. This participant was part of the PPS but not part of the modified Per Protocol Set (N=409).
  participants
    Full Analysis Set | 57 | 56 | 45 | 49 | 54 | 56 | 317
    Per Protocol Set: number analyzed (Participants) | 67 | 68 | 71 | 67 | 68 | 69 | 410
    Per Protocol Set | 46 | 48 | 38 | 39 | 45 | 48 | 264
    modified Per Protocol Set: number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69 | 409
    modified Per Protocol Set | 45 | 48 | 38 | 39 | 45 | 48 | 263

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Double-blind Treatment in Sitting Diastolic Blood Pressure at Trough
Description: Participants had their blood pressure measured at the study site using the BpTRU® device. The BpTRU® is an automatic unattended office blood pressure measurement device. Six measurements, at rest, per participant per visit were performed. The mean of the last 5 measurements was used for the analysis.
  The absolute change in mean trough sitting diastolic blood pressure (SiDBP) measured by from baseline (i.e., at randomization) to week 8 (Day 56). A negative change indicates a decrease in the diastolic blood pressure from the start of treatment.
Time Frame: Baseline (Day 1) and end of double-blind treatment (Day 56)
Population: Modified Per-protocol set (mPPS). All participants who had a mean trough sitting diastolic blood pressure (SiDBP) at Week-8 of the double-blind treatment period and that did not have any major protocol deviation were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
Number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69
mmHg
  Baseline | 97.5 (5.4) | 97.8 (5.5) | 97.7 (4.3) | 97.8 (4.8) | 98.2 (5.3) | 96.8 (4.6)
  Absolute Change from Baseline to Week 8 | -4.9 (11.1) | -6.3 (8.9) | -9.9 (8.7) | -12.0 (8.2) | -10.0 (7.9) | -8.4 (9.6)
Statistical Analysis 1: Comparison: Placebo vs Aprocitentan 5 mg vs Aprocitentan 10 mg vs Aprocitentan 25 mg vs Aprocitentan 50 mg; Multiple Comparison Procedure-Modeling (MCP-Mod) was used to assess a dose-response across placebo and all aprocitentan doses. The null hypothesis of "no dose-response" was rejected if at least one of the six Multiple Contrast Tests (MCTs) had a multiplicity adjusted p-value <0.05. The analysis was performed using the R-package "DoseFinding" (Bornkamp B, Pinheiro J, Bretz F. Planning and analyzing dose finding experiments. 2016. Available from: cran.r-projects.org/web/packages/DoseFinding.); Test type: Other; p < 0.001, Multiple Comparison Procedure-Modeling
Statistical Analysis 2: Comparison: Placebo vs Aprocitentan 5 mg; Test type: Superiority; p = 0.8117, ANCOVA; with Dunnett correction; LS Mean = -1.31, 95% CI 2-sided [-5.10 to 2.49], Standard Error of Mean 1.548
Statistical Analysis 3: Comparison: Placebo vs Aprocitentan 10 mg; Test type: Superiority; p = 0.0053, ANCOVA; with Dunnett correction; LS Mean = -4.93, 95% CI 2-sided [-8.68 to -1.17], Standard Error of Mean 1.532
Statistical Analysis 4: Comparison: Placebo vs Aprocitentan 25 mg; Test type: Superiority; p < .0001, ANCOVA; with Dunnett correction; LS Mean = -6.99, 95% CI 2-sided [-10.80 to -3.19], Standard Error of Mean 1.554
Statistical Analysis 5: Comparison: Placebo vs Aprocitentan 50 mg; Test type: Superiority; p = 0.0057, ANCOVA; with Dunnett correction; LS Mean = -4.95, 95% CI 2-sided [-8.75 to -1.15], Standard Error of Mean 1.549

2. Secondary Outcome: Change From Baseline to End of Double-blind Treatment in Sitting Systolic Blood Pressure at Trough
Description: Participants had their blood pressure measured at the study site using the BpTRU® device. The BpTRU® is an automatic unattended office blood pressure measurement device. Six measurements, at rest, per participant per visit were performed. The mean of the last 5 measurements was used for the analysis.
  The absolute change in mean trough sitting systolic blood pressure (SiSBP) measured by from baseline (i.e., at randomization) to week 8 (Day 56). A negative change indicates a decrease in the systolic blood pressure from the start of treatment.
Time Frame: Baseline (Day 1) and end of double-blind treatment (Day 56)
Population: Modified Per-protocol set (mPPS). All participants who had a mean trough sitting systolic blood pressure (SiSBP) at Week 8 of the double-blind treatment period and that did not have any major protocol deviation were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
Number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69
mmHg
  Baseline | 149.2 (13.1) | 149.4 (13.9) | 149.8 (12.7) | 151.2 (13.7) | 148.6 (12.8) | 149.8 (14.2)
  Absolute Change from Baseline to Week 8 | -7.7 (18.8) | -10.3 (15.3) | -15.0 (14.5) | -18.5 (15.0) | -15.1 (11.8) | -12.8 (16.0)
Statistical Analysis 1: Comparison: Placebo vs Aprocitentan 5 mg vs Aprocitentan 10 mg vs Aprocitentan 25 mg vs Aprocitentan 50 mg; Multiple Comparison Procedure-Modeling (MCP-Mod) was used to assess a dose-response across placebo and all aprocitentan doses. The null hypothesis of "no dose-response" was rejected if at least one of the six Multiple Contrasts Tests (MCTs) had a multiplicity adjusted p-value <0.05. The analysis was performed using the R-package "DoseFinding" (Bornkamp B, Pinheiro J, Bretz F. Planning and analyzing dose finding experiments. 2016. Available from: cran-rprojects.org/web/packages/DoseFinding.); Test type: Other; p < 0.001, Multiple Comparison Procedure-Modeling
Statistical Analysis 2: Comparison: Placebo vs Aprocitentan 5 mg; Test type: Superiority; p = 0.7071, ANCOVA; with Dunnett correction; LS Mean = -2.45, 95% CI 2-sided [-8.44 to 3.54], Standard Error of Mean 2.445
Statistical Analysis 3: Comparison: Placebo vs Aprocitentan 10 mg; Test type: Superiority; p = 0.0138, ANCOVA; with Dunnett correction; LS Mean = -7.05, 95% CI 2-sided [-12.98 to -1.12], Standard Error of Mean 2.420
Statistical Analysis 4: Comparison: Placebo vs Aprocitentan 25 mg; Test type: Superiority; p = 0.0003, ANCOVA; with Dunnett correction; LS Mean = -9.90, 95% CI 2-sided [-15.92 to -3.88], Standard Error of Mean 2.457
Statistical Analysis 5: Comparison: Placebo vs Aprocitentan 50 mg; Test type: Superiority; p = 0.0077, ANCOVA; with Dunnett correction; LS Mean = -7.58, 95% CI 2-sided [-13.58 to -1.59], Standard Error of Mean 0.0077

3. Secondary Outcome: Control Rates at the End of the Double-blind Treatment Period Based on Trough Sitting Diastolic and Systolic Blood Pressure
Description: Participants had their blood pressure measured at the study site using the BpTRU® device. The BpTRU® is an automatic unattended office blood pressure measurement device. Six measurements, at rest, per participant per visit were performed. The mean of the last 5 measurements was used for the analysis. The Canadian Hypertension Education Program (CHEP) issued guidelines proposing cut-offs of 85 mmHg for diastolic blood pressure and 135 mmHg for systolic blood pressure specifically focusing on measurement by automated office blood pressure measurement. The number of participants at the end of the 8-week treatment period that had values below the protocol and CHEP cut-off values are reported.
  The initial protocol control rates at Week 8 (Day 56) on trough SiDBP are also reported and were defined as a SiDBP of less than 90 mmHg and a SiSBP of less than 140 mmHg.
Time Frame: End of double-blind treatment (Day 56)
Population: Modified Per Protocol Set (mPPS). All participants who had diastolic and systolic blood pressure measurements at Week 8 of the double-blind treatment period and that did not have any major protocol deviation were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
Number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69
Participants
  SiDBP less than 90 mmHg | 22 | 30 | 37 | 43 | 39 | 38
  SiDBP less than 85 mmHg (CHEP) | 17 | 15 | 29 | 29 | 21 | 23
  SiSBP less than 140 mmHg | 34 | 37 | 43 | 44 | 47 | 39
  SiSBP less than 135 mmHg (CHEP) | 24 | 27 | 32 | 38 | 36 | 31

4. Secondary Outcome: Response Rates at End of Double-blind Treatment Period Based on Trough Sitting Diastolic Blood Pressure
Description: Participants had their blood pressure measured at the study site using the BpTRU® device. The BpTRU® is an automatic unattended office blood pressure measurement device. Six measurements, at rest, per participant per visit were performed. The mean of the last 5 measurements was used for the analysis.
  A participant was a responder if the reduction from baseline in mean trough sitting diastolic blood pressure (SiDBP) was 10 mmHg or greater-than 10 mmHg.
Time Frame: Baseline (Day 1) and end of double-blind treatment (Day 56)
Population: Modified Per Protocol Set (mPPS).
Measure: Count of Participants; unit: Participants
Groups:
- Lisinopril 20 mg: 20 mg
  Lisinopril: 20 mg capsules orally o.d. for 8 weeks
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
Number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69
Participants | 21 | 21 | 34 | 40 | 38 | 31

5. Secondary Outcome: Response Rates at End of Double-blind Treatment Period Based on Trough Sitting Systolic Blood Pressure
Description: Participants had their blood pressure measured at the study site using the BpTRU® device. The BpTRU® is an automatic unattended office blood pressure measurement device. Six measurements, at rest, per participant per visit were performed. The mean of the last 5 measurements was used for the analysis.
  A participant was a responder if the reduction from baseline in mean trough sitting systolic blood pressure (SiSBP) was 20 mmHg or greater-than 20 mmHg.
Time Frame: Baseline (Day 1) and end of double-blind treatment (Day 56)
Population: Modified Per Protocol Set (mPPS).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
Number analyzed (Participants) | 66 | 68 | 71 | 67 | 68 | 69
Participants | 16 | 16 | 22 | 28 | 22 | 20

6. Secondary Outcome: Change From Baseline to End of Double-blind Treatment in 24-hour Diastolic and Systolic Ambulatory Blood Pressure Monitoring (ABPM)
Description: Diastolic and systolic ambulatory blood pressure monitoring was performed over a 24-hour period with the ABPM device (Mobil-o-Graph) set to record diastolic and systolic blood pressure at a pre-defined time. Over a 24-hour period 3 measurements per hour during the day and 2 per hour during the night were made. The blood pressure measurements were derived from the area under the diastolic and systolic blood pressure curves and divided by the time span and averaged.
  For ambulatory blood pressure monitoring the baseline was the period from the time of last run-in placebo intake up to the time of the first double-blind treatment intake.
Time Frame: Baseline (Day -1 to Day 1) and end of double-blind treatment (Day 55 and Day 56)
Population: All participants in a treatment group with a full set of ABPM (Ambulatory Blood Pressure Monitoring) values over the 24-hour period at baseline and at Week 8.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
Number analyzed (Participants) | 27 | 36 | 36 | 30 | 33 | 30
mmHg
  Baseline 24-hour mean DBP | 90.46 (10.66) | 90.60 (10.19) | 92.60 (10.92) | 89.28 (9.53) | 91.53 (10.54) | 91.18 (9.48)
  Absolute change in 24-hour mean DBP at Week 8 | -2.49 (5.52) | -3.76 (6.36) | -6.55 (7.04) | -8.86 (7.35) | -5.98 (6.63) | -5.72 (9.12)
  Baseline 24-hour mean SBP | 140.28 (14.2) | 139.90 (15.87) | 144.30 (15.68) | 140.83 (11.23) | 141.28 (14.73) | 143.35 (17.53)
  Absolute change in 24-hour mean SBP at Week 8 | -3.54 (7.46) | -3.16 (10.54) | -7.72 (11.37) | -9.23 (9.92) | -6.07 (8.93) | -7.23 (14.33)

7. Secondary Outcome: Ratio of Group Mean at Trough to Group Mean at Peak for Diastolic Blood Pressure Based on Ambulatory Blood Pressure Monitoring (ABPM)
Description: Ratio of group mean at trough to group mean at peak was calculated from the diastolic ambulatory blood pressure monitoring performed over a 24-hour period with the ABPM device. The trough (the smallest blood pressure reduction) and the peak (the highest blood pressure reduction) ratio show the extent of blood pressure lowering throughout the 24-hour dosing interval in the group.
  The group mean trough (at 20-24 hours) to group mean (at 2-6 hours) peak of diastolic blood pressure were examined to evaluate the extent to which once-daily dosing criteria were met (trough-to-peak values greater than 0.5).
  The ratio is positive if there was a decrease in diastolic blood pressure at both the trough and peak times at the end of treatment (Day 55 to Day 56) when compared to baseline (Day -1 to Day 1).
  For ambulatory blood pressure monitoring the baseline was the period from the time of last run-in placebo intake up to the time of the first double-blind treatment intake.
Time Frame: Baseline (Day -1 to Day 1) and end of double-blind treatment (Day 55 and Day 56)
Population: as for outcome 6
Measure: Number; unit: Ratio of mean at trough to mean at peak
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
Number analyzed (Participants) | 27 | 37 | 36 | 30 | 33 | 30
Ratio of mean at trough to mean at peak | -48.03 | 2.59 | 0.90 | 1.49 | 1.25 | 0.65

8. Other Pre Specified Outcome: Supportive Analysis of Primary Endpoint: Change From Baseline to End of Double-blind Treatment in Sitting Diastolic Blood Pressure at Trough
Description: as for outcome 1
Time Frame: Baseline (Day -1 to Day 1) and end of double-blind treatment (Day 55 and Day 56)
Population: The Full Analysis Set (FAS) includes all participants randomized who had a baseline mean trough SiDBP. Participants were evaluated according to the study treatment they have been assigned to. Missing data was analyzed by LOCF (Last Observation Carried Forward).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
Number analyzed (Participants) | 81 | 79 | 80 | 77 | 77 | 79
mmHg
  Baseline | 98.0 (5.5) | 97.5 (5.3) | 97.7 (4.2) | 98.2 (5.0) | 98.4 (5.3) | 96.9 (4.4)
  Absolute Change from Baseline to Week 8 | -4.2 (11.1) | -5.8 (8.9) | -9.9 (8.4) | -11.7 (7.8) | -9.9 (7.8) | -8.2 (9.7)
Statistical Analysis 1: Comparison: Placebo vs Aprocitentan 5 mg vs Aprocitentan 10 mg vs Aprocitentan 25 mg vs Aprocitentan 50 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Multiple Comparison Procedure-Modeling
Statistical Analysis 2: Comparison: Placebo vs Aprocitentan 5 mg; Test type: Superiority; p = 0.5356, ANCOVA; with Dunnett correction; LS Mean = -1.75, 95% CI 2-sided [-5.19 to 1.69], Standard Error of Mean 1.401
Statistical Analysis 3: Comparison: Placebo vs Aprocitentan 10 mg; Test type: Superiority; p = 0.0001, ANCOVA; with Dunnett correction; LS Mean = -5.82, 95% CI 2-sided [-9.25 to -2.40], Standard Error of Mean 1.396
Statistical Analysis 4: Comparison: Placebo vs Aprocitentan 25 mg; Test type: Superiority; p < .0001, ANCOVA; with Dunnett correction; LS Mean = -7.50, 95% CI 2-sided [-10.96 to -4.04], Standard Error of Mean 1.410
Statistical Analysis 5: Comparison: Placebo vs Aprocitentan 50 mg; Test type: Superiority; p = 0.0003, ANCOVA; with Dunnett correction; LS Mean = -5.65, 95% CI 2-sided [-9.11 to -2.19], Standard Error of Mean 1.410

ADVERSE EVENTS:
Time Frame: Up to 12 weeks after first intake of medication after randomization.
Description: The treatment-emergent adverse events were defined as those adverse events with onset on or after the first day of double-blind study treatment intake up to the last day of double-blind study treatment intake plus 30 days.
Groups:
- Placebo: Participants received placebo orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Aprocitentan 5 mg: Participants received aprocitentan 5 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Aprocitentan 10 mg: Participants received aprocitentan 10 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Aprocitentan 25 mg: Participants received aprocitentan 25 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Aprocitentan 50 mg: Participants received aprocitentan 50 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
- Lisinopril 20 mg: Participants received lisinopril 20 mg orally once daily in the morning for 8 weeks during the double-blind treatment period, followed by a 2-week single-blind placebo washout period, followed by a further two-week follow-up period.
Arm/Group | Placebo | Aprocitentan 5 mg | Aprocitentan 10 mg | Aprocitentan 25 mg | Aprocitentan 50 mg | Lisinopril 20 mg
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82 | 0/82 | 0/82 | 0/81 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82 | 0/82 | 2/82 | 0/81 | 1/81
Other Adverse Events (participants affected / at risk) | 30/82 | 18/82 | 24/82 | 32/82 | 22/81 | 25/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Aprocitentan 5 mg (N=82) | Aprocitentan 10 mg (N=82) | Aprocitentan 25 mg (N=82) | Aprocitentan 50 mg (N=81) | Lisinopril 20 mg (N=81)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Aprocitentan 5 mg (N=82) | Aprocitentan 10 mg (N=82) | Aprocitentan 25 mg (N=82) | Aprocitentan 50 mg (N=81) | Lisinopril 20 mg (N=81)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lens disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vitreous degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Tenderness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 4 (4)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Norovirus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine free increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruxism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition frequency decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mole excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT02603809/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT02603809/SAP_001.pdf